CLINICAL TRIAL: NCT04507152
Title: Effect of Blood Flow Restriction Resistance Training on Muscle Strength and Functional Performance in Frail Older Adults
Brief Title: Blood Flow Restriction Training in Pre-frail and Frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Pei-Yun Lee, Assistant professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-BR-108-111-T
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Frailty
Keywords: Blood flow restriction; Resistance exercise; Frailty
MeSH Terms: conditions — Frailty | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction resistance training (Experimental)
  Interventions: Other: Blood flow restriction resistance training
- Resistance training (Active Comparator)
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Blood flow restriction resistance training — The participants will carry weights and perform certain resistance exercises, such as step-up, sit-to-stand, and tip-toe-standing. The experimental group will execute the training with blood flow restriction.
  Arms: Blood flow restriction resistance training
Other: Resistance training — The participants will carry weights and perform certain resistance exercises, such as step-up, sit-to-stand, and tip-toe-standing. The control group will execute the training without blood flow restriction.
  Arms: Resistance training

SUMMARY:
Frailty is most often defined as a syndrome of physiological decline in late life, characterized by marked vulnerability to adverse health outcomes. Intervention such as exercise, especially resistance exercise, has proven to be effective to improve frail condition in the elderly in the previous literature. However, blood flow restriction (BFR) training, a new resistance exercise training method, need merely lower resistance power and shorter training duration compared with traditional resistance exercise. Previous researches also demonstrated BFR can increase muscle mass and muscle strength in the healthy elderly but the effect of BFR training on the pre-frail or frail elderly is unknown. The aim of this study will test the effect of BFR training on muscle strength and functional performance in pre-frail or frail elderly. Participants aged over 60 years old with clinical frailty score between 3 to 5 will be recruited. Participants will be assigned to two groups using randomized block design with BFR training and control group. Structured questionnaire and physical function measurement will be used to assess the pre-intervention condition and outcome of different interventions. The participants will be assessed before training (pre-test), 3 weeks after training, and 6 weeks after training (post-test), and followed up at one and three months after training. Physical function measurement will include hand grip, muscle mass over trunk and extremity, muscle strength of lower extremity, gait speed and timed up and go test. Two-way repeated measures analysis of variance will be used to test the pre-test, 3-week, post-test and follow-ups difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 60 years old
* Fried frailty index fulfill 1-2 criteria
* Able to walk 6 meters independently
* Able to understand and follow ≥ 3 instructions

Exclusion Criteria:

* Severe hypertension (>180/110mmHg)
* Peripheral neuropathy
* History of deep-vein thrombosis (DVT)
* Cardiovascular diseases (i.e. Heart failure NYHA Classification III or IV, myocardial infarction, pulmonary hypertension, coronary artery stenosis)
* Neuromuscular diseases (i.e. Stroke, Parkinsons' disease)
* History of resisted exercise training program within the last 6 months before screening

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Change of muscle strength of the lower extremities | Before training, 3 and 6 weeks after training, and one and two months follow-ups
  Bilateral hip flexors, knee extensors, ankle dorsiflexors and ankle plantarflexors
Change of 30 seconds sit to stand | Before training, 3 and 6 weeks after training, and one and two months follow-ups
  30 seconds sit to stand
Change of timed-up-and-go test | Before training, 3 and 6 weeks after training, and one and two months follow-ups
  Timed-up-and-go test

SECONDARY OUTCOMES:
Change of one-repetition maximum | Before training, 3 and 6 weeks after training, and one and two months follow-ups
  One-repetition maximum of step-ups
Change of muscle mass | Before training, 3 and 6 weeks after training, and one and two months follow-ups
  Muscle mass of the upper and lower extremities and trunk
Change of hand grip | Before training, 3 and 6 weeks after training, and one and two months follow-ups
  Bilateral hand grip strength
Change of physical activity level | Before training, 3 and 6 weeks after training, and one and two months follow-ups
  The International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No